CLINICAL TRIAL: NCT00857909
Title: The Effect of Amiloride and Spironolactone Measured on Cardiovascular and Kidney Related Variables in Healthy Subjects in a Double-blinded, Randomised, Placebo-controlled, Cross-over Study
Brief Title: The Effect of Amiloride and Spironolactone in Healthy Persons
Acronym: SPAS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Erling Bjerregaard Pedersen/ Dr. Med, Medical Research Department
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MED.RES:HOS:SKM.02.2009
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2011-07

CONDITIONS: High Blood Pressure
MeSH Terms: conditions — Hypertension | interventions — Amiloride; Spironolactone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Randomisation 1 (Active Comparator): Amiloride 5 mg twice daily for 28 days, later compared with spironolactone and placebo
  Interventions: Drug: Amiloride; Drug: Placebo and spironolactone
- Randomisation 2 (Active Comparator): Spironolactone 25 mg twice daily, to be compared with placebo and amiloride
  Interventions: Drug: Spironolactone
- Placebo (Placebo Comparator): calcium tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amiloride — 1 tablet twice a day
  Arms: Randomisation 1
Drug: Spironolactone — 1 tablet twice a day
  Arms: Randomisation 2
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Placebo and spironolactone — 5mg twice daily
  Arms: Randomisation 1
Drug: Spironolactone — 25mg twice daily
  Arms: Randomisation 2

SUMMARY:
This study will investigate whether retaining potassium in the body will lead to changes in blood pressure and changes in blood and urine samples.

DETAILED DESCRIPTION:
The purpose is to measure the effect of amiloride and spironolactone on:

1. Renal function (GFR, u-AQP2, u-ENaCβ, u-cAMP, u-PGE2, CH20, FENa, FEK),
2. Pulsbewave velocity, augmentation index and central blood pressure,
3. Vasoactive hormones (PRC, AngII, Aldo, AVP, ANP, BNP and Endot), and
4. Ambulatory blood pressure

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-smokers

Exclusion Criteria:

* Smoking
* Under medical treatment

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, Prof, Principal Investigator — Regional Hospital Holstebro
Locations (1):
- Medical Research, Holstebro, Denmark